CLINICAL TRIAL: NCT01262417
Title: Evaluationof the Efficiency of a Resorbable Barrier Membrane for the Prevention of Abdominal and Peri-hepatic Adhesion in Patients With Colorectal Cancer Requiring Two-stage Surgery for the Resection of Hepatic Metastases
Brief Title: Resorbable Barrier for the Prevention of Abdominal and Peri-hepatic Adhesion Formation
Acronym: SEPRAC2T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Zora ABDELBOST, Centre Léon Bérard, 28 rue Laënnec, 69373, Lyon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SEPRAC2T
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; two stage surgery for the resection of hepatic metastases; resorbable barrier membrane; abdominal and peri-hepatic adhesion
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Seprafilm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- - Seprafilm group (Experimental): patients receiving resorbable barrier membrane during the first surgery
  Interventions: Procedure: - use of resorbable membrane Seprafilm
- - No-treatment control group (Other): patients without seprafilm barrier during the first surgery
  Interventions: Procedure: without resorbable barrier (seprafilm)

INTERVENTIONS:
Procedure: - use of resorbable membrane Seprafilm — use of resorbable membrane during the first surgery for the resection of hepatic metastases, 1 to 4 membranes should be used around the liver
  Other Names: use of Seprafilm after the resction of hepatic metastases
  Arms: - Seprafilm group
Procedure: without resorbable barrier (seprafilm) — non use of resorbable membrane during the first surgery for the resection of hepatic metastases
  Other Names: resection of hepatic metastases
  Arms: - No-treatment control group

SUMMARY:
The purpose of this study is to evaluate the efficiency of a resorbable barrier membrane for the prevention of abdominal and peri-hepatic adhesion in patients with colorectal cancer requiring two-stage surgery for the resection of hepatic metastases.

Eligible patients will be randomly assigned to one of 2 arms:

* Seprafilm group (receiving resorbable barrier membrane during the first surgery)
* No-treatment control group (without seprafilm barrier during the first surgery)

The primary objective is to establish, in patients with colorectal cancer requiring two-stage surgery for the resection of hepatic metastases, the efficiency of a resorbable barrier membrane (Seprafilm) for limiting abdominal and peri-hepatic adhesion during the second operation.

This study is a prospective multicentric phase II, controlled, randomized and non comparative trial.

A total of 60 patients will be enrolled: 45 will receive Seprafilm whereas 15 will be assigned to the no-treatment control group. The inclusion period should be approximately 18 months. The follow up period after the second surgery will be 3 years.

DETAILED DESCRIPTION:
The secondary objectives of the study are:

During and after the 1st surgical procedure To evaluate immediate complications (during surgery), early complications (during post-surgery hospitalization) and late complications (between 1st and 2nd surgeries) in relation with operating procedure and use of resorbable membrane.

During and after the 2nd surgical procedure

* To evaluate abdominal and peri-hepatic adhesion (at the site of the 1st surgery), with qualitative and quantitative description.
* To evaluate intestinal adhesion (in the small intestine), with quantitative description.
* To evaluate immediate complications (during surgery), early complications (during post-surgery hospitalization) and late complications (in the month following the intervention) in relation with operating procedure.
* To evaluate post-operative rehabilitation
* To assess tumour evolution in patients over a period of 3 years after the 2nd surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged ≥ 18 years
* Colorectal cancer with synchronous or metachronous hepatic metastases
* Patients requiring two-stage surgery with laparotomy for the resection of hepatic metastases
* The 2 operations should be scheduled in the same centre
* The 2 operations should be scheduled at an interval of 1 to 6 months
* Patient affiliated with social security
* Patient able to read and write French
* Written, voluntary, informed consent

Exclusion Criteria:

* Patient with previous hepatic or biliary surgery through supra-umbilical incision (except biliary surgery with laparotomy more than 6 months previously)
* Patient with previous major surgery except colorectal surgery for resection of primitive tumour
* Metastasis removable in one surgical procedure
* Non resectable metastasis
* Follow-up impossible for social, geographical, familial or psychological reasons
* Patient deprived of freedom
* Patient enrolled in another experimental surgery trial
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
abdominal and peri-hepatic adhesion during the second operation | Time to liberate liver (t0: incision and t1: liberation)

SECONDARY OUTCOMES:
immediate complications during the first surgical procedure in relation with operating procedure and use of resorbable membrane | during the surgery
early complications (after the 1st surgical procedure)in relation with operating procedure and use of resorbable membrane | during post-surgery hospitalization
late complications (after the 1st surgical procedure)in relation with operating procedure and use of resorbable membrane | between 1st and 2nd surgeries (2 operations should be scheduled at an interval of 1 to 6 months)
abdominal and peri-hepatic adhesion (at the site of the 1st surgery), with qualitative and quantitative description | at the beginning of the 2nd surgical procedure
intestinal adhesion (in the small intestine), with quantitative description | at the beginning of the second surgical procedure
immediate complications in relation with operating procedure. | during the 2nd surgical procedure
early complications (after 2ng operation) in relation with operating procedure. | during post-surgery hospitalization
late complications in relation with operating procedure. | in the month following the 2nd intervention
post-operative rehabilitation | during post-surgery hospitalization
tumour evolution in patients | over a period of 3 years after the 2nd surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michel Rivoire, MD, Principal Investigator — Centre Léon Bérard, Lyon
Locations (17):
- France (17):
  - Institut Bergonié, Bordeaux
  - Hôpital Antoine Béclère, Clamart
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHU Grenoble, Grenoble
  - Centre Hospitalier Lyon Sud, Lyon
  - Centre Léon Bérard, Lyon
  - Hôpital de La Croix Rousse, Lyon
  - CHU La conception, Marseille
  - Institut Paoli Calmettes, Marseille
  - Centre Val d'Aurelle Paul Lamarque, Montpellier
  - Centre Alexis Vautrin, Nancy
  - Hôpital de Brabois CHU, Nancy
  - CHU Nice-Hôpital de l'Archet II, Nice
  - Hôpital Cochin, Paris
  - Hôpital Charles Nicolle - CHU Rouen, Rouen
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Weibel MA, Majno G. Peritoneal adhesions and their relation to abdominal surgery. A postmortem study. Am J Surg. 1973 Sep;126(3):345-53. doi: 10.1016/s0002-9610(73)80123-0. No abstract available. PMID 4580750
- [Background] Adam R, Laurent A, Azoulay D, Castaing D, Bismuth H. Two-stage hepatectomy: A planned strategy to treat irresectable liver tumors. Ann Surg. 2000 Dec;232(6):777-85. doi: 10.1097/00000658-200012000-00006. PMID 11088072
- [Background] Jaeck D, Oussoultzoglou E, Rosso E, Greget M, Weber JC, Bachellier P. A two-stage hepatectomy procedure combined with portal vein embolization to achieve curative resection for initially unresectable multiple and bilobar colorectal liver metastases. Ann Surg. 2004 Dec;240(6):1037-49; discussion 1049-51. doi: 10.1097/01.sla.0000145965.86383.89. PMID 15570209
- [Background] Ellis H, Moran BJ, Thompson JN, Parker MC, Wilson MS, Menzies D, McGuire A, Lower AM, Hawthorn RJ, O'Brien F, Buchan S, Crowe AM. Adhesion-related hospital readmissions after abdominal and pelvic surgery: a retrospective cohort study. Lancet. 1999 May 1;353(9163):1476-80. doi: 10.1016/S0140-6736(98)09337-4. PMID 10232313
- [Background] Beck DE, Opelka FG, Bailey HR, Rauh SM, Pashos CL. Incidence of small-bowel obstruction and adhesiolysis after open colorectal and general surgery. Dis Colon Rectum. 1999 Feb;42(2):241-8. doi: 10.1007/BF02237135. Erratum In: Dis Colon Rectum 1999 May;42(5):578. PMID 10211502
- [Background] Diamond MP, Freeman ML. Clinical implications of postsurgical adhesions. Hum Reprod Update. 2001 Nov-Dec;7(6):567-76. doi: 10.1093/humupd/7.6.567. PMID 11727865
- [Background] Ray NF, Denton WG, Thamer M, Henderson SC, Perry S. Abdominal adhesiolysis: inpatient care and expenditures in the United States in 1994. J Am Coll Surg. 1998 Jan;186(1):1-9. doi: 10.1016/s1072-7515(97)00127-0. PMID 9449594
- [Background] Lower AM, Hawthorn RJ, Ellis H, O'Brien F, Buchan S, Crowe AM. The impact of adhesions on hospital readmissions over ten years after 8849 open gynaecological operations: an assessment from the Surgical and Clinical Adhesions Research Study. BJOG. 2000 Jul;107(7):855-62. doi: 10.1111/j.1471-0528.2000.tb11083.x. PMID 10901556
- [Background] Lower AM, Hawthorn RJ, Clark D, Boyd JH, Finlayson AR, Knight AD, Crowe AM; Surgical and Clinical Research (SCAR) Group. Adhesion-related readmissions following gynaecological laparoscopy or laparotomy in Scotland: an epidemiological study of 24 046 patients. Hum Reprod. 2004 Aug;19(8):1877-85. doi: 10.1093/humrep/deh321. Epub 2004 Jun 3. PMID 15178659
- [Background] Parker MC, Ellis H, Moran BJ, Thompson JN, Wilson MS, Menzies D, McGuire A, Lower AM, Hawthorn RJ, O'Briena F, Buchan S, Crowe AM. Postoperative adhesions: ten-year follow-up of 12,584 patients undergoing lower abdominal surgery. Dis Colon Rectum. 2001 Jun;44(6):822-29; discussion 829-30. doi: 10.1007/BF02234701. PMID 11391142
- [Background] Parker MC. Epidemiology of adhesions: the burden. Hosp Med. 2004 Jun;65(6):330-6. doi: 10.12968/hosp.2004.65.6.13729. PMID 15222206
- [Background] Bristow RE, Montz FJ. Prevention of adhesion formation after radical oophorectomy using a sodium hyaluronate-carboxymethylcellulose (HA-CMC) barrier. Gynecol Oncol. 2005 Nov;99(2):301-8. doi: 10.1016/j.ygyno.2005.06.057. Epub 2005 Aug 8. PMID 16085295
- [Background] Bristow RE, Santillan A, Diaz-Montes TP, Gardner GJ, Giuntoli RL 2nd, Peeler ST. Prevention of adhesion formation after radical hysterectomy using a sodium hyaluronate-carboxymethylcellulose (HA-CMC) barrier: a cost-effectiveness analysis. Gynecol Oncol. 2007 Mar;104(3):739-46. doi: 10.1016/j.ygyno.2006.09.029. Epub 2006 Nov 13. PMID 17097723
- [Background] Duron JJ. [Post-operative bowel obstruction. Part 2: Mechanical post-operative small bowel obstruction by bands and adhesions]. J Chir (Paris). 2003 Dec;140(6):325-34. French. PMID 14978440
- [Background] Duron JJ. [Post-operative bowel obstruction. Part 1: Intraperitoneal bands and adhesions--causes and prevention]. J Chir (Paris). 2003 Sep;140(4):211-9. French. PMID 13679770
- [Background] Cuervas-Mons V, Rimola A, Van Thiel DH, Gavaler JS, Schade RR, Starzl TE. Does previous abdominal surgery alter the outcome of pediatric patients subjected to orthotopic liver transplantation? Gastroenterology. 1986 Apr;90(4):853-7. doi: 10.1016/0016-5085(86)90860-7. PMID 3512356
- [Background] Sandler AD, Azarow KS, Superina RA. The impact of a previous Kasai procedure on liver transplantation for biliary atresia. J Pediatr Surg. 1997 Mar;32(3):416-9. doi: 10.1016/s0022-3468(97)90594-7. PMID 9094006
- [Background] Ong TH. Prevention of intraabdominal adhesions in Kasai portoenterostomy. J Pediatr Surg. 2001 Nov;36(11):1613-4. doi: 10.1053/jpsu.2001.27930. PMID 11685684
- [Background] Jaeck D, Bachellier P, Guiguet M, Boudjema K, Vaillant JC, Balladur P, Nordlinger B. Long-term survival following resection of colorectal hepatic metastases. Association Francaise de Chirurgie. Br J Surg. 1997 Jul;84(7):977-80. doi: 10.1002/bjs.1800840719. PMID 9240140
- [Background] Rivoire M; ANAES. [Can initially non-respectable hepatic metastases be made resectable?]. Gastroenterol Clin Biol. 2003 Mar;27 Spec No 2:B18-9, B88-104. No abstract available. French. PMID 12637875
- [Background] Al-Jaroudi D, Tulandi T. Adhesion prevention in gynecologic surgery. Obstet Gynecol Surv. 2004 May;59(5):360-7. doi: 10.1097/00006254-200405000-00024. PMID 15097797
- [Background] Beck DE, Cohen Z, Fleshman JW, Kaufman HS, van Goor H, Wolff BG; Adhesion Study Group Steering Committee. A prospective, randomized, multicenter, controlled study of the safety of Seprafilm adhesion barrier in abdominopelvic surgery of the intestine. Dis Colon Rectum. 2003 Oct;46(10):1310-9. doi: 10.1007/s10350-004-6739-2. PMID 14530667
- [Background] Becker JM, Dayton MT, Fazio VW, Beck DE, Stryker SJ, Wexner SD, Wolff BG, Roberts PL, Smith LE, Sweeney SA, Moore M. Prevention of postoperative abdominal adhesions by a sodium hyaluronate-based bioresorbable membrane: a prospective, randomized, double-blind multicenter study. J Am Coll Surg. 1996 Oct;183(4):297-306. PMID 8843257
- [Background] Diamond MP. Reduction of adhesions after uterine myomectomy by Seprafilm membrane (HAL-F): a blinded, prospective, randomized, multicenter clinical study. Seprafilm Adhesion Study Group. Fertil Steril. 1996 Dec;66(6):904-10. PMID 8941053
- [Background] Salum MR, Lam DT, Wexner SD, Pikarsky A, Baig MK, Weiss EG, Nogueras JJ, Singh JJ. Does limited placement of bioresorbable membrane of modified sodium hyaluronate and carboxymethylcellulose (Seprafilm) have possible short-term beneficial impact? Dis Colon Rectum. 2001 May;44(5):706-12. doi: 10.1007/BF02234571. PMID 11357033
- [Background] Tang CL, Seow-Choen F, Fook-Chong S, Eu KW. Bioresorbable adhesion barrier facilitates early closure of the defunctioning ileostomy after rectal excision: a prospective, randomized trial. Dis Colon Rectum. 2003 Sep;46(9):1200-7. doi: 10.1007/s10350-004-6716-9. PMID 12972964
- [Background] Vrijland WW, Tseng LN, Eijkman HJ, Hop WC, Jakimowicz JJ, Leguit P, Stassen LP, Swank DJ, Haverlag R, Bonjer HJ, Jeekel H. Fewer intraperitoneal adhesions with use of hyaluronic acid-carboxymethylcellulose membrane: a randomized clinical trial. Ann Surg. 2002 Feb;235(2):193-9. doi: 10.1097/00000658-200202000-00006. PMID 11807358
- [Background] Tingstedt B, Isaksson K, Andersson E, Andersson R. Prevention of abdominal adhesions--present state and what's beyond the horizon? Eur Surg Res. 2007;39(5):259-68. doi: 10.1159/000102591. Epub 2007 May 10. PMID 17495476
- [Background] Oikonomakis I, Wexner SD, Gervaz P, You SY, Secic M, Giamundo P. Seprafilm: a retrospective preliminary evaluation of the impact on short-term oncologic outcome in colorectal cancer. Dis Colon Rectum. 2002 Oct;45(10):1376-80. doi: 10.1007/s10350-004-6428-1. PMID 12394438
- [Background] Kusunoki M, Ikeuchi H, Yanagi H, Noda M, Tonouchi H, Mohri Y, Uchida K, Inoue Y, Kobayashi M, Miki C, Yamamura T. Bioresorbable hyaluronate-carboxymethylcellulose membrane (Seprafilm) in surgery for rectal carcinoma: a prospective randomized clinical trial. Surg Today. 2005;35(11):940-5. doi: 10.1007/s00595-005-3061-0. PMID 16249848
- [Background] Wieand HS. Randomized phase II trials: what does randomization gain? J Clin Oncol. 2005 Mar 20;23(9):1794-5. doi: 10.1200/JCO.2005.10.956. Epub 2005 Feb 7. No abstract available. PMID 15699476
- [Background] Dixon WJ, Massey FJ. Introduction to statistical analysis. 4th Edition McGraw-Hill, 1983; 80-5.
- [Background] Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. J Am Stat Assoc 1958; 53: 457-81.
- [Derived] Dupre A, Lefranc A, Buc E, Delpero JR, Quenet F, Passot G, Evrard S, Rivoire M. Use of bioresorbable membranes to reduce abdominal and perihepatic adhesions in 2-stage hepatectomy of liver metastases from colorectal cancer: results of a prospective, randomized controlled phase II trial. Ann Surg. 2013 Jul;258(1):30-6. doi: 10.1097/SLA.0b013e3182854949. PMID 23426344